CLINICAL TRIAL: NCT01941251
Title: Navigated Alpha Frequency Transcranial Magnetic Stimulation (αTMS) in Treatment-resistant Schizophrenia
Brief Title: Navigated αTMS in Treatment-resistant Schizophrenia
Acronym: nTMS_NS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Niuvanniemi Hospital (Other)
Responsible Party: Principal Investigator, Heli Tuppurainen, MD, PhD, Niuvanniemi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 932012
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; Schizophrenia; Schizoaffective Disorder; Treatment; Negative Symptoms; Positive Symptoms; TMS; rTMS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigated individualized αTMS (Active Comparator): navigated Transcranial Magnetic Stimulation
  Interventions: Device: navigated Transcranial Magnetic Stimulation
- Sham TMS (Sham Comparator): navigated Transcranial Magnetic Stimulation using sham coil
  Interventions: Device: navigated Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: navigated Transcranial Magnetic Stimulation — * individualized α frequency
  * left DLPFC 110% motor threshold (MT)
  * 13-15 sessions for 3 weeks
  Other Names: TMS; rTMS
  Arms: Navigated individualized αTMS
Device: navigated Transcranial Magnetic Stimulation — - placebo treatment: sham coil
  Other Names: TMS; rTMS
  Arms: Sham TMS

SUMMARY:
Since 1990s, stimulation of prefrontal cortex (PFC) has shown therapeutic effects on auditory hallucinations as well as negative symptoms of schizophrenia. However, previous studies have reported mixed or negative results. Majority of the repetitive transcranial magnetic stimulation (rTMS) studies to date has set the target of cortical stimulation based on scalp site. Recently introduced method, navigated transcranial magnetic stimulation (nTMS) integrates the individual MRI data, and thus allows more precise targeting on brain cortical regions enhancing the efficacy of rTMS. Previous EEG studies have suggested reduced alpha band activity in patients with schizophrenia. Some recent studies using alpha (α) EEG guided TMS for treating positive and negative symptoms of schizophrenia have demonstrated promising results.

The aim of the study is to investigate the efficacy of navigated individualized αTMS in treatment-resistant patients with schizophrenia. Approximately fifty patients with DSM-IV schizophrenia will be enrolled in this randomized, double-blind, sham-controlled study. The patients will receive 13 - 15 session of αTMS to the left dorsolateral prefrontal cortex (DLPFC), as adjunctive therapy, for 3 weeks. We assess patients via the Positive and Negative Syndrome Scale (PANSS), Clinical Global Impression (CGI) and neurocognitive test battery at baseline, 5 days after and 3 months after treatment. Serum and plasma levels of brain derived neurotrophic factor (BDNF) are assayed at pre and post treatment weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male righthanded inpatients, 18 to 64 years of age
* The diagnosis of Schizophrenia or Schizoaffective Disorder according to DSM-IV
* Capacity and willingness to give informed consent
* Patient is treatment-resistant, CGI-S 4 or more
* Patient is not requiring a change in antipsychotic medication 2 weeks prior to or during treatment
* No foreseeable changes in patient's smoking habits during treatment

Exclusion Criteria:

* Serious somatic illness
* Progressive neurological illness, recent brain damage (less than 3 months ago) or sequela of serious brain damage
* Unstable epilepsy
* Electro convulsive therapy (ECT) less than 3 months prior to treatment

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | at baseline,5 days after treatment, 3 months after treatment
  change in PANSS total, positive, negative and general psychopathology sum score

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement scale (CGI-I) | at 5 days after treatment, 3 months after treatment
  change in patient's illness relative to baseline state
Neuropsychology test battery | at baseline, 5 days after treatment, 3 months after treatment
  Neuropsychology test battery consists of 6 tests for measuring neurocognitive function.

OTHER OUTCOMES:
plasma and serum levels of Brain Derived Neurotrophic Factor (P-/S-BDNF) | at baseline, 1 week after treatment
  change in P-/S-BDNF levels

CONTACTS AND LOCATIONS:
Overall Officials: Heli Tuppurainen, MD, PhD, Principal Investigator — Niuvanniemi Hospital
Locations (1):
- Niuvanniemi Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Tuppurainen H, Maatta S, Kononen M, Julkunen P, Kautiainen H, Hyvarinen S, Vaurio O, Joensuu M, Vanhanen M, Aho-Mustonen K, Mervaala E, Tiihonen J. Navigated and individual alpha-peak-frequency-guided transcranial magnetic stimulation in male patients with treatment-refractory schizophrenia. J Psychiatry Neurosci. 2024 Mar 1;49(2):E87-E95. doi: 10.1503/jpn.230063. Print 2024 Jan-Feb. PMID 38428970